CLINICAL TRIAL: NCT04363320
Title: Fostering MAT Use in Justice Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: George Mason University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019-1473; 3U2CDA050097-01S1 (NIH); 20200548 (Other: WIRB protocol number); A195010 (Other: UW Madison); ENGR/CHESS PROGRAM (Other: UW Madison)
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Opioid-use Disorder; Recidivism
Keywords: MOUD; OUD; Justice Populations; Jails; ECHO; NIATx; Inter-agency
MeSH Terms: conditions — Opioid-Related Disorders; Recidivism

STUDY DESIGN:
Intervention Model Description: The proposed study will implement a cluster randomized block design where staff are nested within sites. The community-based provider sites and jails will be grouped into homogeneous blocks and then randomly assigned into 2x2 factorial design for each block. The forty-eights sites will be assigned to one of four study arms using a matching strategy within the blocks that groups four jail-clinic combination together prior to randomization. Each jail and cognitive behavioral (CB) treatment provider (or clinic) in these combinations will be treated as a site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-Dose NIATx Coaching & ECHO (Experimental): * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * 12 monthly (one-hour) coaching calls with Change Leader/Team
  * Prescribers participate in 12 monthly (one-hour) scheduled video conference calls
  Interventions: Behavioral: NIATx Coaching; Behavioral: ECHO
- Low-Dose NIATx Coaching & ECHO (Experimental): * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * Four (one-hour) coaching calls at months 1, 4, 8, and 12 with Change Leader/Team
  * Prescribers participate in 12 monthly (one-hour) scheduled video conference calls
  Interventions: Behavioral: NIATx Coaching; Behavioral: ECHO
- High-Dose NIATx Coaching & No ECHO (Experimental): * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * 12 monthly (one-hour) coaching calls with Change Leader/Team
  Interventions: Behavioral: NIATx Coaching
- Low-Dose NIATx Coaching & No ECHO (Experimental): * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * Four (one-hour) coaching calls at months 1, 4, 8, and 12 with Change Leader/Team
  Interventions: Behavioral: NIATx Coaching

INTERVENTIONS:
Behavioral: NIATx Coaching — NIATx framework provides each participating site with a NIATx Coach who is an expert in MOUD implementation and organizational change and will help the organization adopt, implement, and increase the use of MOUD. Coaches help the sites think through key issues, offer process improvement training, and suggest changes.
Behavioral: ECHO — The ECHO model connects MOUD prescribers and experts with primary care providers and medical teams to promote high-quality MOUD practices. ECHO is provided monthly through videoconferences. Experienced MOUD prescribers address topics such as counseling strategies, urine test interpretation, and transitioning from buprenorphine, naltrexone and methadone.
  Other Names: Extension for Community Healthcare Outcomes
  Arms: High-Dose NIATx Coaching & ECHO; Low-Dose NIATx Coaching & ECHO

SUMMARY:
The grant will test two timely and successful evidence-based implementation practices, NIATx Coaching and ECHO, with jail/community-based healthcare providers to increase medication assisted treatment (MAT) use with justice populations.

DETAILED DESCRIPTION:
In this trial, the investigators will test two implementation interventions being applied to medications for opioid use disorder (MOUD) dissemination and implementation in justice settings for justice-involved populations: NIATx Coaching and the Extension for Community Healthcare Outcomes (ECHO) model. NIATx Coaches provide expertise in MOUD implementation and organizational change to help treatment organizations and staff make, sustain, and spread MOUD. The ECHO platform focuses only on the provider side by connecting the primary care provider with expert MOUD prescribers to promote high-quality MOUD practices. This will be the first trial that assesses the comparative effectiveness of these approaches overall, and in justice settings.

The trial will be conducted with a combination of 48 jails and community-based organizations that treat individuals with opioid use disorders (OUDs) post-incarceration. Sites will be randomly assigned to one of four study arms, with 12 sites in each arm: High-Dose Coaching/ECHO, Low-Dose Coaching/ECHO, High-Dose Coaching/No ECHO, and Low-Dose Coaching/No ECHO. The intervention period will be over a 12-month span with an additional 12-months for sustainability.

ELIGIBILITY:
Site Inclusion Criteria:

* Have an interest in embedding or increasing the use of MOUD within their site.
* Have the funds to pay for medications for the duration of the study (24 months); whether it be from grants, insurance or private pay.
* Sites agree to implement or continue to use at least one medication, although they will be encouraged to offer more than one medication.
* Have leadership support at all levels.
* Agree to provide data described in the MOU or Information Sheet.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, PhD, Principal Investigator — University of Wisconsin, Madison; Faye Taxman, PhD, Principal Investigator — George Mason University
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Molfenter T, Vechinski J, Kim JS, Zhang J, Meng L, Tveit J, Madden L, Taxman FS. Assessing the comparative effectiveness of ECHO and coaching implementation strategies in a jail/provider MOUD implementation trial. Implement Sci. 2025 Feb 3;20(1):7. doi: 10.1186/s13012-025-01419-6. PMID 39901259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 48 sites were recruited, 38 (25 jails & 13 Community based treatment provider (CBTP) sites completed the study (sites per intervention listed in the participant flow). Consenting Participants are staff at the sites who provided data, including counts of people prescribed medications for opioid use disorder (MOUD) at their sites (see outcome measures for this data).
Units Other Than Participants: Sites
Groups:
- High-Dose NIATx Coaching & ECHO: * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * 12 monthly (one-hour) coaching calls with Change Leader/Team
  * Prescribers participate in 12 monthly (one-hour) scheduled video conference calls
  NIATx Coaching: NIATx framework provides each participating site with a NIATx Coach who is an expert in MOUD implementation and organizational change and will help the organization adopt, implement, and increase the use of MOUD. Coaches help the sites think through key issues, offer process improvement training, and suggest changes.
  ECHO: The ECHO model connects MOUD prescribers and experts with primary care providers and medical teams to promote high-quality MOUD practices. ECHO is provided monthly through videoconferences. Experienced MOUD prescribers address topics such as counseling strategies, urine test interpretation, and transitioning from buprenorphine, naltrexone and methadone.
- Low-Dose NIATx Coaching & ECHO: * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * Four (one-hour) coaching calls at months 1, 4, 8, and 12 with Change Leader/Team
  * Prescribers participate in 12 monthly (one-hour) scheduled video conference calls
  NIATx Coaching: NIATx framework provides each participating site with a NIATx Coach who is an expert in MOUD implementation and organizational change and will help the organization adopt, implement, and increase the use of MOUD. Coaches help the sites think through key issues, offer process improvement training, and suggest changes.
  ECHO: The ECHO model connects MOUD prescribers and experts with primary care providers and medical teams to promote high-quality MOUD practices. ECHO is provided monthly through videoconferences. Experienced MOUD prescribers address topics such as counseling strategies, urine test interpretation, and transitioning from buprenorphine, naltrexone and methadone.
- High-Dose NIATx Coaching & No ECHO: * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * 12 monthly (one-hour) coaching calls with Change Leader/Team
  NIATx Coaching: NIATx framework provides each participating site with a NIATx Coach who is an expert in MOUD implementation and organizational change and will help the organization adopt, implement, and increase the use of MOUD. Coaches help the sites think through key issues, offer process improvement training, and suggest changes.
- Low-Dose NIATx Coaching & No ECHO: * Four-hour, Virtual Kick-Off Meeting split into two days with Study Team & Coaches
  * Four (one-hour) coaching calls at months 1, 4, 8, and 12 with Change Leader/Team
  NIATx Coaching: NIATx framework provides each participating site with a NIATx Coach who is an expert in MOUD implementation and organizational change and will help the organization adopt, implement, and increase the use of MOUD. Coaches help the sites think through key issues, offer process improvement training, and suggest changes.
Period: Overall Study
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Started (Staff were consented at sites.) | 78; 14 Sites | 65; 11 Sites | 60; 10 Sites | 53; 13 Sites
Completed (Reasons for sites dropping included change in leadership (new leadership not interested in participating), lack of referrals from the jail, or doors closed due to lack loss of funding.) | 35; 9 Sites | 23; 10 Sites | 35; 9 Sites | 24; 10 Sites
Not Completed | 43; 5 Sites | 42; 1 Sites | 25; 1 Sites | 29; 3 Sites
Not completed — Lost to Follow-up | 43 | 42 | 24 | 29
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The overall number analyzed includes the count of staff participants consented. The overall number of units analyzed is the number of sites that started the study.
Units Other Than Participants: Sites Starting Study
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO | Total
Number analyzed (Participants) | 78 | 65 | 60 | 53 | 256
Number analyzed (Sites Starting Study) | 14 | 11 | 10 | 13 | 48
Age, Continuous [Mean (Full Range); unit: years] | 46 [24 to 68] | 42 [22 to 74] | 46 [24 to 74] | 46 [24 to 76] | 46 [22 to 76]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 45 | 39 | 32 | 30 | 146
  Male | 23 | 22 | 27 | 20 | 92
  Unknown | 10 | 4 | 1 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 9 | 0 | 1 | 15
  Not Hispanic or Latino | 64 | 52 | 59 | 49 | 224
  Unknown or Not Reported | 9 | 4 | 1 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 0 | 0 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 1 | 4
  Black or African American | 17 | 2 | 10 | 7 | 36
  White | 37 | 50 | 44 | 38 | 169
  More than one race | 4 | 5 | 2 | 0 | 11
  Unknown or Not Reported | 11 | 7 | 4 | 4 | 26
Region of Enrollment [Number; unit: participants]
  United States | 78 | 65 | 60 | 53 | 256
Geographic Location of Sites [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics.
  Sites Starting Study
    Rural | 3 | 5 | 4 | 3 | 15
    Suburban | 1 | 3 | 3 | 6 | 13
    Urban | 10 | 3 | 3 | 4 | 20
Gender Served [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics.
  Sites Starting Study
    Male only | 0 | 1 | 0 | 0 | 1
    Female only | 0 | 0 | 0 | 0 | 0
    Both | 14 | 10 | 10 | 13 | 47
Average Daily Population (Jails only) [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics for Jails only.
  Sites Starting Study
    number analyzed (Participants) | 51 | 42 | 50 | 37 | 180
    number analyzed (Sites Starting Study) | 8 | 7 | 7 | 7 | 29
    less than 100 | 1 | 3 | 2 | 0 | 6
    101-250 | 1 | 3 | 1 | 5 | 10
    251-500 | 2 | 0 | 3 | 1 | 6
    greater than 500 | 4 | 1 | 1 | 1 | 7
Average Monthly OUD Intakes (CBTP) [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics for CBTP only.
  Sites Starting Study
    number analyzed (Participants) | 27 | 23 | 10 | 16 | 76
    number analyzed (Sites Starting Study) | 6 | 4 | 3 | 6 | 19
    less than 50 | 3 | 0 | 1 | 3 | 7
    51-200 | 0 | 2 | 1 | 0 | 3
    201-500 | 0 | 0 | 1 | 0 | 1
    greater than 500 | 0 | 0 | 0 | 1 | 1
    unknown | 3 | 2 | 0 | 2 | 7
Type of Healthcare Model at Jails [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics at Jails only.
  Sites Starting Study
    number analyzed (Participants) | 51 | 42 | 50 | 37 | 180
    number analyzed (Sites Starting Study) | 8 | 7 | 7 | 7 | 29
    Direct | 3 | 2 | 1 | 1 | 7
    Contracted | 4 | 4 | 1 | 4 | 13
    Hybrid | 1 | 1 | 5 | 2 | 9
CBTP Arrangements with Jails [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics CBTP only.
  Sites Starting Study
    number analyzed (Participants) | 27 | 23 | 10 | 16 | 76
    number analyzed (Sites Starting Study) | 6 | 4 | 3 | 6 | 19
    Joint Staffings | 3 | 1 | 1 | 2 | 7
    Shared Written Agreements | 3 | 2 | 3 | 3 | 11
    Electronic Health Record Access | 2 | 0 | 2 | 0 | 4
    Referral Processes | 3 | 3 | 3 | 4 | 13
MOUD Offered at Baseline [Count of Units; unit: Sites Starting Study] — Population: Data applies to site characteristics.
  Sites Starting Study
    Buprenorphine/Naloxone | 10 | 8 | 7 | 11 | 36
    Naltrexone (injectable) | 8 | 10 | 5 | 7 | 30
    Naltrexone (oral) | 6 | 4 | 6 | 6 | 22
    Methadone | 7 | 3 | 6 | 2 | 18
    No MOUD | 0 | 0 | 1 | 0 | 1
    Unknown | 1 | 0 | 0 | 1 | 2
Type of Study Site [Count of Units; unit: Sites Starting Study]
  Jails | 8 | 7 | 7 | 7 | 29
  Community Based Treatment Providers | 6 | 4 | 3 | 6 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of New Eligible Justice Involved Persons Initiated With MOUD Per Month: Intervention Phase
Description: The intervention reach will be measured using data gathered through organization monthly tracking sheets to track MOUD use. 'Involved persons' include those who are initiated onto any MOUD (buprenorphine, extended-release injectable naltrexone, or methadone) and engaged with MOUD use.
Time Frame: baseline to 12 months
Population: The Overall Number of Participants Analyzed reported are justice involved individuals staff (who were not consented and enrolled). Staff (consented participants) collected counts of justice involved individuals with various MOUD from their sites. Not all sites provided all three forms of medication at all times. Due to lack of tracking systems in the jail, some sites were only able to provide one of the two monthly counts.
Measure: Mean (Standard Deviation); unit: New Justice Involved Persons per month
Units Other Than Participants: sites
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 4572 | 256 | 569 | 1908
Number analyzed (sites) | 14 | 11 | 10 | 13
New Justice Involved Persons per month
  Methadone: number analyzed (sites) | 9 | 10 | 6 | 9
  Methadone | 20.36 (51.31) | 0.55 (1.57) | 4.47 (9.63) | 2.03 (5.57)
  Buprenorphine: number analyzed (sites) | 9 | 8 | 4 | 8
  Buprenorphine | 21.79 (28.5) | 3.00 (4.05) | 5.01 (2.98) | 17.43 (25.56)
  Naltrexone: number analyzed (sites) | 9 | 8 | 6 | 9
  Naltrexone | 0.19 (0.28) | 0.33 (0.42) | 0.44 (0.86) | 1.37 (2.05)
Statistical Analysis 1: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Combined MOUD) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.002, Mixed Models Analysis — a prior threshold 0.05; Slope = 0.538, Standard Deviation 0.169 — Slope is per month
Statistical Analysis 2: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Buprenorphine) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.0008, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.38, Standard Deviation 0.113 — Slope is per month
Statistical Analysis 3: Comparison: High-Dose NIATx Coaching & No ECHO; Change in new patient counts (Methadone) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.111, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.207, Standard Deviation 0.129 — Slope is per month
Statistical Analysis 4: Comparison: Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Naltrexone) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.235, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.017, Standard Deviation 0.014 — Slope is per month

2. Primary Outcome: Mean Number of New Eligible Justice Involved Persons Initiated With MOUD Per Month: Sustainability Phase
Description: as for outcome 1
Time Frame: 13 months, 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: New Justice Involved Persons per month
Units Other Than Participants: sites
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 6345 | 240 | 542 | 3022
Number analyzed (sites) | 14 | 11 | 10 | 13
New Justice Involved Persons per month
  Methadone: number analyzed (sites) | 9 | 8 | 4 | 8
  Methadone | 28.29 (75.24) | 0.01 (0.03) | 4.67 (6.6) | 2.41 (6.31)
  Buprenorphine: number analyzed (sites) | 9 | 6 | 3 | 7
  Buprenorphine | 30.37 (35.77) | 3.3 (4.4) | 7.89 (3.18) | 32.32 (60.72)
  Naltrexone: number analyzed (sites) | 9 | 6 | 4 | 8
  Naltrexone | 0.09 (0.13) | 1.32 (1.59) | 0.71 (0.79) | 0.79 (1.01)
Statistical Analysis 1: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Combined MOUD) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.485, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.153, Standard Deviation 0.218 — Slope is per month
Statistical Analysis 2: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new Justice Involved Person counts (Buprenorphine) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.0008, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.642, Standard Deviation 0.19 — Slope is per month
Statistical Analysis 3: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Methadone) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.015, Mixed Models Analysis — a priori threshold: 0.05; Slope = -0.377, Standard Deviation 0.154 — Slope is per month
Statistical Analysis 4: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in new patient counts (Naltrexone) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.241, Mixed Models Analysis — a priori threshold: 0.05; Slope = -0.02, Standard Deviation 0.017 — Slope is per month

3. Primary Outcome: Mean Total Number of Eligible Justice Involved Persons on MOUD Per Month: Intervention Phase
Description: as for outcome 1
Time Frame: baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Justice Involved Persons per month
Units Other Than Participants: sites
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 19120 | 8588 | 9025 | 6263
Number analyzed (sites) | 14 | 11 | 10 | 13
Justice Involved Persons per month
  Methadone: number analyzed (sites) | 9 | 9 | 8 | 9
  Methadone | 98.73 (216.36) | 0.08 (0.35) | 56.58 (158.40) | 0.94 (1.80)
  Buprenorphine: number analyzed (sites) | 8 | 6 | 7 | 9
  Buprenorphine | 104.07 (145.32) | 117.62 (190.42) | 36.50 (45.29) | 60.57 (105.31)
  Naltrexone: number analyzed (sites) | 8 | 7 | 8 | 9
  Naltrexone | 0.24 (0.34) | 2.60 (5.29) | 5.81 (15.04) | 3.21 (6.16)
Statistical Analysis 1: Comparison: High-Dose NIATx Coaching & ECHO; Change in census patient counts (Combined MOUD) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.00002, Mixed Models Analysis — a priori threshold: 0.05; Slope = 1.912, Standard Deviation 0.438 — Slope is per month
Statistical Analysis 2: Comparison: Low-Dose NIATx Coaching & ECHO; Change in census patient counts (Buprenorphine) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.00004, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.855, Standard Deviation 0.206 — Slope is per month
Statistical Analysis 3: Comparison: High-Dose NIATx Coaching & No ECHO; Change in census patient counts (Methadone) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.118, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.322, Standard Deviation 0.206 — Slope is per month
Statistical Analysis 4: Comparison: Low-Dose NIATx Coaching & No ECHO; Change in census patient counts (Naltrexone) for Intervention Phase (from baseline to 12 months); Test type: Superiority; p = 0.020, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.073, Standard Deviation 0.031 — Slope is per month

4. Primary Outcome: Mean Total Number of Eligible Justice Involved Persons on MOUD Per Month: Sustainability Phase
Description: as for outcome 1
Time Frame: 13 months to 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Justice Involved Persons per month
Units Other Than Participants: sites
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 24145 | 5799 | 9489 | 8041
Number analyzed (sites) | 14 | 11 | 10 | 13
Justice Involved Persons per month
  Methadone: number analyzed (sites) | 9 | 8 | 6 | 8
  Methadone | 110.19 (219.28) | 0.01 (0.03) | 77.22 (183.37) | 1.96 (3.71)
  Buprenorphine: number analyzed (sites) | 8 | 5 | 6 | 8
  Buprenorphine | 127.32 (177.17) | 154.78 (227.42) | 43.71 (43.31) | 78.24 (136.17)
  Naltrexone: number analyzed (sites) | 8 | 4 | 6 | 8
  Naltrexone | 0.22 (0.31) | 1.67 (1.56) | 10.86 (18.72) | 3.7 (6.44)
Statistical Analysis 1: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in census patient counts (Combined MOUD) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.045, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.617, Standard Deviation 0.307 — Slope is per month
Statistical Analysis 2: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in census patient counts (Buprenorphine) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.000002, Mixed Models Analysis — a priori threshold: 0.05; Slope = 1.103, Standard Deviation 0.229 — Slope is per month
Statistical Analysis 3: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in census patient counts (Methadone) for Sustainability Phase (13 to 24 months); Test type: Superiority; p = 0.076, Mixed Models Analysis — a priori threshold: 0.05; Slope = -0.387, Standard Deviation 0.218 — Slope is per month
Statistical Analysis 4: Comparison: High-Dose NIATx Coaching & ECHO vs Low-Dose NIATx Coaching & ECHO vs High-Dose NIATx Coaching & No ECHO vs Low-Dose NIATx Coaching & No ECHO; Change in census patient counts (Naltrexone) for Sustainability Phase (from 13 to 24 months); Test type: Superiority; p = 0.019, Mixed Models Analysis — a priori threshold: 0.05; Slope = 0.086, Standard Deviation 0.036 — Slope is per month

5. Primary Outcome: Change in Number of Prescribers Using MOUD
Description: The adoption of each intervention will be in part measured by tracking the number of prescribers using MOUD at each time point.
Time Frame: baseline, 12 months, 24 months
Population: Data was not collected for this outcome. This outcome was determined to not be a key variable at study start and should have been removed from the protocol. It was apparent from listening to sites that increasing the number of prescribers was not a goal as they were already encountering high turnover rates and staffing.
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: MOUD Sustainability Measured Using the Program Sustainability Assessment Tool
Description: The maintenance of the intervention (MOUD Sustainability) will be measured using the Program Sustainability Assessment Tool included in the Staff Survey at three points during the study (baseline, 12-months & 24-months) to determine if likelihood of sustainability increases as study progresses. This tool has a total possible range of scores from 0-63 with higher scores indicating increased sustainability of the intervention.
Time Frame: baseline, 12 months, 24 months
Population: Number of participants and sites included in data analysis changed through study conduct.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: sites
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 78 | 65 | 60 | 53
Number analyzed (sites) | 14 | 11 | 10 | 13
score on a scale
  baseline | 44.79487 (17.88808) | 43.75385 (15.68342) | 43.16667 (14.61386) | 43.96226 (12.7701)
  12 months: number analyzed (Participants) | 42 | 28 | 45 | 21
  12 months: number analyzed (sites) | 10 | 10 | 10 | 10
  12 months | 50.71429 (8.827025) | 50.78571 (8.252304) | 45.95556 (10.73642) | 51.61905 (10.70736)
  24 months: number analyzed (Participants) | 35 | 23 | 35 | 24
  24 months: number analyzed (sites) | 9 | 10 | 9 | 10
  24 months | 51.51429 (13.18504) | 49.30435 (8.704413) | 48.37143 (11.95847) | 53.70833 (14.0077)

7. Other Pre Specified Outcome: NIATx Fidelity
Description: Assess fidelity to the NIATx implementation strategies at two points during the study using a 10-item measure with scores ranging from 0-40 with higher scores indicating stronger fidelity of the intervention.
Time Frame: 12 months, 24 months
Population: Number of participants included in data analysis changed through study conduct.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
Number analyzed (Participants) | 78 | 65 | 60 | 53
score on a scale
  12 months: number analyzed (Participants) | 42 | 28 | 45 | 21
  12 months | 24.2381 (6.449842) | 25.39286 (4.474945) | 24.11111 (6.544332) | 24.71429 (5.917287)
  24 months: number analyzed (Participants) | 35 | 23 | 35 | 24
  24 months | 24.57143 (5.494841) | 23.13043 (4.07101) | 24.62857 (7.272372) | 27.16667 (6.112472)

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | High-Dose NIATx Coaching & ECHO | Low-Dose NIATx Coaching & ECHO | High-Dose NIATx Coaching & No ECHO | Low-Dose NIATx Coaching & No ECHO
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/65 | 1/60 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/65 | 0/60 | 0/53
Other Adverse Events (participants affected / at risk) | 0/78 | 0/65 | 0/60 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/20/NCT04363320/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT04363320/ICF_001.pdf